CLINICAL TRIAL: NCT04765969
Title: Determination of Factors Related With Daily Living Activities in Severe COPD
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, Vice-dean of Faculty of Health Sciences (PhD, PT), Halic University
Other Study IDs: ssaka1
Record Dates: First submitted 2020-03-16; First posted 2021-02-23 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: COPD
Keywords: COPD; Activities of Daily Living
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe COPD patients: GOLD C and D group patients

SUMMARY:
The main purpose of chronic obstructive pulmonary disease (COPD) rehabilitation applications is to increase the functional capacity of the patients and improve the quality of life in daily living activities (ADL). Therefore, the investigators planned the study to determine the influence of ADL and related factors in severe COPD.

GOLD C and D COPD patients admitted to Bezmialem Vakif University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Pulmonary Rehabilitation Application and Research Laboratory will be included in this study on a voluntary basis. Individuals who have experienced exacerbations of COPD in the last 6 weeks, have comorbidities affecting ambulation and have cognitive impairment will be excluded. Physical and sociodemographic characteristics of all participants will be recorded. Spirometric measurement will used to evaluate pulmonary functions, London Chest Activities Scale (LCADL) will used to evaluate daily living activities, six minute walking test (6MWT) will used to evaluate functional capacity, and mouth pressure will measured to evaluate respiratory muscle strength. (MIP: maximal inspiratory pressure, MEP: maximal expiratory pressure). Saint George Respiratory Questionnaire (SGRQ) for assessing quality of life, International Physical Activity Questionnaire (IPAQ) for assessing physical activity, COPD Assessment Test (CAT) for symptom assessment, and Hospital Anxiety and Depression Scale (HAD) for anxiety and depression assessment will be applied. SPSS 22.0 package program will be used in statistical analysis. For descriptive statistics, mean ± standard deviation values will be calculated and Pearson correlation test will be used in correlation analysis. p <0.05 will be the level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary function tests (PFT) value of FEV₁ / FVC <70%,
* Being in GOLD III-IV groups,
* Being over 18 years old,
* Being able to read and to understand the spoken language.

Exclusion Criteria:

* subjects have had COPD exacerbation in the last six weeks,
* having comorbidities affecting ambulation and
* cognitive disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD subjects who were referred to the Bezmialem Vakıf University
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Activities of daily living | 6 months
  The LCADL Scale is going to used to assess dyspnea resulting from ADL . It consists of a total of 15 items within four domains: personal care (4 items), domestic (6 items), physical (2 items), and leisure (3 items). Each item is graded from 0 to 5 with higher scores indicating more difficulty performing ADL. The scale can be evaluated as total score, domain scores, and item scores. The maximum total score is 75. There is also a single question that assesses to what degree dyspnea perception affects daily life in general. This item is answered by selecting one of three responses: 'a lot', 'a little', or 'not at all'

SECONDARY OUTCOMES:
Pulmonary Function Test | 6 months
  Spirometer is performed according to the American Thoracic Society (ATS) guidelines in Bezmialem University PFT Laboratory with Zan-100 spire (nSpire Health GmbH, Oberthulba, Germany). FVC (l), FEV₁(l), FEV1(%), FEV₁/FVC (%) were recorded.
FEV1 (liter) | 6 months
  This is the amount of air with pulmonary function test that the patient can force out of their lungs in one second.
FEV1 (%-percentage) | 6 months
  This is the percentage of air with pulmonary function test that the patient can force out of their lungs in one second.
FVC (liter) | 6 months
  This is the greatest total amount of air patient can forcefully breathe out after breathing in as deeply as possible.
FEV1/FVC (percentage) | 6 months
  The FEV1/FVC ratio is a number that represents the percentage of patient lung capacity patient is able to exhale in one second.
Inspiratory muscle test | 6 months
  Maximal inspiratory pressure (MIP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).
Functional capacity | 6 months
  Functional capacity is going to assessed with the 6 minute walk test (6MWT) according to the guideline of ATS .
Symptoms | 6 months
  For the symptom burden of COPD, COPD Assessment Test (CAT) is going to used. It consists of eight items, each presented as a semantic 6-point differential scale, providing a score out of 40 indicating the impact of the disease
Physical activity | 6 months
  It provides information about time spent on walking, moderate to severe activities. Time spent in sitting is considered as a separate question. The calculation of the total score of the short form includes the sum of walking, moderate intensity activity, and duration (minutes) and frequency (days) of intensive activity.
Expiratory muscle test | 6 months
  Maximal expiratory pressure (MEP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).

OTHER OUTCOMES:
Health related quality of life assessment | 6 months
  For the assessment of quality of life, Saint George's Respiratory Questionnaire (SGRQ) is going to used. The SGRQ is a 76-item pulmonary disease-specific health related quality of life (HRQL) questionnaire with well-demonstrated reliability and validity in subjects with pulmonary diseases. The SGRQ results are grouped into 3 domains (symptoms, activity, and impacts) and a total score. Scores range from 0 to 100, with a lower score indicating better pulmonary-specific HRQL.
Anxiety and depression | 6 months
  Anxiety and depression is going to assessed with Hospital Anxiety and Depression Scale (HADS). The HADS consists of seven items for anxiety (HADS-A) and seven items for depression (HADS-D). The items are scored on a four-point scale from zero (not present) to three (considerable)

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our clinical datas' are not available for sharig considering ethical problems.

REFERENCES:
- [Result] Ozsoy I, Ozcan Kahraman B, Acar S, Ozalevli S, Akkoclu A, Savci S. Factors Influencing Activities of Daily Living in Subjects With COPD. Respir Care. 2019 Feb;64(2):189-195. doi: 10.4187/respcare.05938. Epub 2018 Nov 6. PMID 30401755
- [Result] Kapella MC, Larson JL, Covey MK, Alex CG. Functional performance in chronic obstructive pulmonary disease declines with time. Med Sci Sports Exerc. 2011 Feb;43(2):218-24. doi: 10.1249/MSS.0b013e3181eb6024. PMID 20543752